CLINICAL TRIAL: NCT05921721
Title: Does the EOS Imaging System Improve Assessment of the Hip in Individuals Aged 13 Years and Over Compared to CT?
Brief Title: Can EOS Hip Imaging Replace CT Hip Scans?
Acronym: EOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheffield Children's NHS Foundation Trust (Other)
Collaborators: EOS imaging Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SCH-2653
Record Dates: First submitted 2023-06-06; First posted 2023-06-27 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Femoroacetabular Impingement; Hip Dysplasia
MeSH Terms: conditions — Femoracetabular Impingement; Hip Dislocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EOS imaging system (Experimental): Participants will undergo CT and EOS imaging pre- and post- operatively. The EOS is being compared to the reference method CT scan.
  Interventions: Device: EOS

INTERVENTIONS:
Device: EOS — This modality simultaneously captures biplanar radiographs (anteroposterior and lateral images) through the whole-body slot scanning with patients in standing position with ultralow irradiation

SUMMARY:
The orientation of the femoral neck in relation to the coronal or transcondylar axis of the distal femur is known as the femoral version. It is categorised as femoral anteversion when the femoral neck axis is anteriorly rotated in relation to transcondylar axis, while femoral head axis is anterior in relation to the femur coronal plane; or femoral retroversion when the femoral head-neck axis points are posterior to the femoral coronal plane.

Some studies suggest that conventional radiography cannot adequately measure femoral version, and should be avoided in favour of more precise methods using computed tomography (CT) scanning. CT imaging is currently the reference method for measuring femoral version. However, its clinical use is limited by issues such as high levels of radiation exposure, which can adversely affect patients, especially children. Magnetic resonance imaging (MRI) is considered an alternative for measuring femoral version; however, it is expensive, time consuming and subject to motion artifacts. The associated costs and risks of MRI increase when anaesthesia is needed for the examination. The EOS imaging system could provide an alternative to the previously mentioned techniques. It uses lower doses of irradiation and the sterEOS software allows the production of 3D images.

This study aims to compare the accuracy of the EOS imaging system with CT for the measurement of hip parameters in individuals aged 13 years and older. In addition, this study aims to correlate EOS and CT parameters with gait analysis and compare the ability of EOS and CT to predict gait abnormalities.

DETAILED DESCRIPTION:
The average range of anteversion at birth is from 30 to 40 degrees. These values reduce with growth, remaining in the10 to 15-degree range for most adults. Nevertheless, these values can be significantly different between populations or contralateral sides. Altered femoral version can affect the normal function and even stability of the hip and knee joints, so that it must be considered in the clinical assessment of cases involving femoral fractures, torsional alignment, slipped capital femoral epiphysis and Legg-Calve-Perthes disease. Femoral version can be evaluated by clinical investigation or radiographic assessment.

Imaging examinations play an important role in the evaluation of femoral version prior to surgical interventions. However, some studies suggest that conventional radiography cannot adequately measure femoral version. CT imaging is currently the reference method for measuring femoral version. However, its clinical use is limited by issues such as high levels of radiation exposure, which can adversely affect patients, especially children. Magnetic resonance imaging (MRI) is considered an alternative for measuring femoral version; however, it is expensive, time consuming and subject to motion artifacts. The associated costs and risks increase when anaesthesia is needed for the examination. The EOS imaging system provides an alternative to the previously mentioned techniques. It uses lower doses of irradiation and the sterEOS software allows the production of 3D images. The EOS system can measure the torsional alignment of the lower limbs with 4 to 30 times less irradiation than a CT scan. Prior studies measuring femoral version using both EOS and CT have found a high correlation between the results of these techniques.

Acetabular morphology and 3D orientation are important factors to be considered prior to orthopaedic surgery. Acetabular orientation is known to vary between genders as women have more anteverted acetabula than men, as well as a larger inclination angle. For hip preservation surgery, the most promising technique for the treatment of dysplasia in adolescents and young adults is peri-acetabular osteotomy (PAO). The benefits of PAO in the treatment of hip joint pathology are discussed in more detail and have been assessed either morphologically using MRI or functionally, by performing post-operative gait analysis.

The EOS imaging system with 3D sterEOS software can produce 3D reconstructions of the acetabulum with 30-fold lower irradiation of patients compared to CT and 10-fold lower irradiation compared to chest radiographs. The innovation behind the EOS system earned its inventor a Nobel prize in physics (particle detection). This modality simultaneously captures biplanar radiographs (anteroposterior and lateral images) through the whole-body slot scanning with patients in standing position with ultralow irradiation. 3D reconstructions of the individual skeleton can be performed from these captured radiographs using sterEOS software. 2D and 3D EOS skeletal images are produced with similar volume and size to 1:1 scale, so that vertebral and spinal angles and lengths of lower limbs and other variable parameters can be measured accurately. The advantage is that sterEOS 3D reconstructions can be useful for evaluating rotational disorders of joints and lower limbs horizontally. The EOS system can acquire 3D information of individuals in standing, sitting and squatting positions.

The EOS system has the advantage of allowing for 3D reconstructions of hip/pelvic parameters with lower irradiation than CT scans. This allows for the identification of underlying deformities while exposing patients to lower radiation dose. It would seem that the EOS system has potential to replace CT as the investigation of choice for assessing hip morphology.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged 13 years and older who are considered eligible to undergo periacetabular osteotomy (PAO).
2. Symptomatic dysplasia (Severin grade II or III) or femoroacetabular impingement.
3. Skeletal maturity, defined on pelvic radiographs by closure of the triradiate cartilage.
4. Absence of subluxation (Severin grade I-III).

Exclusion Criteria:

1. Obvious joint incongruency.
2. Loss of sphericity (Severin IV or above).
3. Evidence of moderate or severe arthritis (Tonnis 2 or above).

Ages: 13 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of EOS | 18 months
  Diagnostic accuracy of the EOS imaging system compared to CT for measuring native hip/pelvic parameters in individuals aged 13 years and older
Inter- and intraobserver reliability of EOS | 18 months
  Inter- and intraobserver reliability of the EOS imaging system compared to CT for measuring native hip/pelvic parameters in individuals aged 13 years and older

SECONDARY OUTCOMES:
Predictive power of EOS | 18 months
  Correlation of pre- and post-operative hip measurements from EOS and CT to predict disturbances in gait and quality of life at 6 and 18 months post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Amaka Offiah, Principal Investigator — University of Sheffield

IPD SHARING:
Plan to Share IPD: No